CLINICAL TRIAL: NCT00046371
Title: Open-Label, Phase II Trial of Immunological Response Rate, Safety, and Tolerability of THERATOPE® Vaccine in Subjects With Metastatic Breast Cancer Undergoing Treatment With Aromatase Inhibitors or Faslodex®
Brief Title: Safety and Immunological Response Rate Study of THERATOPE® Vaccine in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncothyreon Canada Inc. (Industry)
Purpose: Treatment
Other Study IDs: STn-BR-105
Record Dates: First submitted 2002-09-27; First posted 2002-10-10 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Breast Neoplasms
Keywords: Cancer Vaccines; Aromatase; Receptors, Estrogen; Receptors, Progesterone
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: THERATOPE® vaccine

SUMMARY:
The purpose of this study is to examine the immunological response rate to administration of the THERATOPE® vaccine in women with stable metastatic breast cancer who are being treated with aromatase inhibitors or Faslodex® and who do not require chemotherapy.

Post-menopausal women on aromatase inhibitors or Faslodex® alone and pre-menopausal women on aromatase inhibitors plus luteinising hormone-releasing hormone (LH/RH)-agonist may be eligible to be enrolled.

Patients must not have had radiotherapy or major surgery within four (4) weeks prior to entering the study.

Information about the safety and tolerability of administration of the THERATOPE® vaccine will also be gathered during the course of the study.

ELIGIBILITY:
Inclusion Criteria

* Histopathologically confirmed breast cancer
* Documented Stage IV disease
* Estrogen and/or progesterone-receptor positive
* Stable disease on aromatase inhibitor or Faslodex® treatment begun at least 12 weeks prior to enrolment
* Performance status, ECOG = 0 or 1
* Life expectancy > 12 weeks
* History of freedom from progression for at least 6 months following surgery with a curative intent or for at least 6 months during adjuvant chemotherapy, adjuvant radiotherapy or adjuvant hormonal therapy such as tamoxifen/toremifene treatment
* No radiotherapy or major surgery within 4 weeks prior to enrolment

Exclusion Criteria

* Pregnant or lactating
* Known brain metastasis
* Bone marrow involvement as the only site of metastasis
* First line chemotherapy for Stage IV disease
* Past or current cancer other than breast cancer, except for curatively treated basal cell cancer or in situ cancer of the cervix with no evidence of disease
* Autoimmune disease, e. g., type I juvenile onset diabetes mellitus, antibody positive rheumatoid arthritis, Grave's disease, lupus, Crohn's disease, IBD, Hashimoto's thyroiditis
* Known intercurrent infections (including HBV or HCV) or immunosuppression [human immunodeficiency virus (HIV) or other conditions] or clinical evidence of these conditions
* Other significant active infection
* Pleural effusions and/or ascites requiring paracentesis every 2 weeks or more frequently
* Splenectomy
* Concurrent treatment with chemotherapeutic agents other than low-dose cyclophosphamide used in this study
* Treatment with interferons (IFNs), cytokines, systemic steroids or other biologicals within 4 weeks prior to enrolment
* Receipt of another investigational drug within 30 days of enrolment
* Known allergy to shellfish
* Known allergy to soy beans or soy products
* Known hypersensitivity to polysorbate 80
* Known hypersensitivity to the study drugs
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Berkeley, California
  - San Francisco, California
  - Santa Monica, California
  - Jacksonville, Florida
  - Plantation, Florida
  - Port Saint Lucie, Florida
  - Chicago, Illinois
  - Des Moines, Iowa
  - Billings, Montana
  - Morristown, New Jersey
  - Gastonia, North Carolina
  - Hickory, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Houston, Texas
  - Norfolk, Virginia
  - Richmond, Virginia